CLINICAL TRIAL: NCT00482196
Title: To Study Different Levels of MK0493 for Safety, Efficacy, and Tolerability in Obese Patients (0493-017)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0493-017; 2007_577
Record Dates: First submitted 2007-06-01; First posted 2007-06-05 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — N-1-(2-(1-(tert-butyl-4-(2,4-difluorophenyl)pyrrolidin-3-yl)-5-chlorophenyl)ethyl)acetamide

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0493

SUMMARY:
To study different doses of MK0493 for safety, efficacy and tolerability in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 21 and 65 years of age

Exclusion Criteria:

* HIV positive as determined by medical history
* Patient is pregnant, lactating or plans to become pregnant
* Patient has undergone surgical treatment for obesity
* Patient has undergone a surgical procedure within 4 weeks prior to Visit 1 or plans to undergo a surgical procedure during the study
* Patient plans to consume more than 2 glasses of grapefruit juice per day during the study
* Patient has participated in another clinical study (involving an investigational drug) within 3 months prior to restudy screening

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2005-07; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Krishna R, Gumbiner B, Stevens C, Musser B, Mallick M, Suryawanshi S, Maganti L, Zhu H, Han TH, Scherer L, Simpson B, Cosgrove D, Gottesdiener K, Amatruda J, Rolls BJ, Blundell J, Bray GA, Fujioka K, Heymsfield SB, Wagner JA, Herman GA. Potent and selective agonism of the melanocortin receptor 4 with MK-0493 does not induce weight loss in obese human subjects: energy intake predicts lack of weight loss efficacy. Clin Pharmacol Ther. 2009 Dec;86(6):659-66. doi: 10.1038/clpt.2009.167. Epub 2009 Sep 9. PMID 19741604